CLINICAL TRIAL: NCT02866643
Title: Labor and Delivery Implant Insertion: A Randomized Controlled Trial
Acronym: LADII
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Kate Ayers Shaw, Clinical Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-38505
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-06

CONDITIONS: Postpartum Contraception; Family Planning
Keywords: contraceptive implant; postpartum contraception; breastfeeding and contraception
MeSH Terms: conditions — Breast Feeding | interventions — etonogestrel; Contraceptive Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Delivery Room Insertion (Experimental): Participants who randomize to this arm will receive the contraceptive implant in the Labor and Delivery room (0-2 hours following delivery).
  Interventions: Drug: Etonogestrel-Immediate
- Postpartum Insertion (Active Comparator): Participants who randomize to this arm will receive the contraceptive implant in the postpartum ward room before discharge (24-48 hours following delivery).
  Interventions: Drug: Etonogestrel-Delayed

INTERVENTIONS:
Drug: Etonogestrel-Immediate — The investigational intervention will be to insert the contraceptive implant immediately postpartum in the delivery room insertion (0-2 hours following delivery).
  Other Names: Nexplanon; Contraceptive Implant
  Arms: Delivery Room Insertion
Drug: Etonogestrel-Delayed — The investigational intervention will be to insert the contraceptive implant 24-48 hours following delivery.
  Other Names: Nexplanon; Contraceptive Implant
  Arms: Postpartum Insertion

SUMMARY:
A barrier to initiating progestin contraceptives in the early postpartum period is the concern of interference with breastfeeding, specifically lactogenesis. In this trial, the investigators aim to describe the effects of immediate insertion of the contraceptive implant on breastfeeding. The investigators seek to examine the time to lactogenesis with immediate post-delivery insertion in delivery room versus insertion of a contraceptive implant in the postpartum ward prior to medical discharge. For this study, 82 consenting women will be randomized to immediate implant insertion (0-2 hours following delivery) in the delivery room or insertion of the implant following delivery in postpartum room and prior to medical discharge (24-48 hours following delivery).

Participants complete a questionnaire that asks questions about breastfeeding continuation, supplementation, duration, and exclusivity. This questionnaire also includes questions about contraceptive continuation, patient satisfaction with implant, pregnancy, and postpartum care visits.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are patients of the Stanford University Obstetrics service
* Pregnant women who delivery a healthy infant, regardless of gestational age.
* Intend to breastfeed
* Desire the contraceptive implant as their method of contraception
* Agree to be randomized to delivery room vs. postpartum ward insertion

Exclusion Criteria:

* Not English or Spanish speaking
* Allergy or Contraindication to contraceptive implant.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kate A Shaw, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Obstetrics--Lucile Packard Children's Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Finer LB, Zolna MR. Declines in Unintended Pregnancy in the United States, 2008-2011. N Engl J Med. 2016 Mar 3;374(9):843-52. doi: 10.1056/NEJMsa1506575. PMID 26962904
- [Background] Zhu BP. Effect of interpregnancy interval on birth outcomes: findings from three recent US studies. Int J Gynaecol Obstet. 2005 Apr;89 Suppl 1:S25-33. doi: 10.1016/j.ijgo.2004.08.002. PMID 15820365
- [Background] Zhu BP, Rolfs RT, Nangle BE, Horan JM. Effect of the interval between pregnancies on perinatal outcomes. N Engl J Med. 1999 Feb 25;340(8):589-94. doi: 10.1056/NEJM199902253400801. PMID 10029642
- [Background] Mayer JP. Unintended childbearing, maternal beliefs, and delay of prenatal care. Birth. 1997 Dec;24(4):247-52. doi: 10.1111/j.1523-536x.1997.tb00598.x. PMID 9460316
- [Background] Heller R, Cameron S, Briggs R, Forson N, Glasier A. Postpartum contraception: a missed opportunity to prevent unintended pregnancy and short inter-pregnancy intervals. J Fam Plann Reprod Health Care. 2016 Apr;42(2):93-8. doi: 10.1136/jfprhc-2014-101165. Epub 2015 Dec 8. PMID 26645197
- [Background] Speroff L, Mishell DR Jr. The postpartum visit: it's time for a change in order to optimally initiate contraception. Contraception. 2008 Aug;78(2):90-8. doi: 10.1016/j.contraception.2008.04.005. Epub 2008 Jun 12. No abstract available. PMID 18672108
- [Background] Centers for Disease Control and Prevention (CDC). Postpartum care visits--11 states and New York City, 2004. MMWR Morb Mortal Wkly Rep. 2007 Dec 21;56(50):1312-6. PMID 18097343
- [Background] Gariepy AM, Duffy JY, Xu X. Cost-Effectiveness of Immediate Compared With Delayed Postpartum Etonogestrel Implant Insertion. Obstet Gynecol. 2015 Jul;126(1):47-55. doi: 10.1097/AOG.0000000000000907. PMID 26241255
- [Background] Centers for Disease Control and Prevention (CDC). Contraceptive use among postpartum women - 12 states and New York City, 2004-2006. MMWR Morb Mortal Wkly Rep. 2009 Aug 7;58(30):821-6. PMID 19661855
- [Background] Centers for Disease Control and Prevention (CDC). Update to CDC's U.S. Medical Eligibility Criteria for Contraceptive Use, 2010: revised recommendations for the use of contraceptive methods during the postpartum period. MMWR Morb Mortal Wkly Rep. 2011 Jul 8;60(26):878-83. PMID 21734635
- [Background] Medical Eligibility Criteria for Contraceptive Use. 5th edition. Geneva: World Health Organization; 2015. Available from http://www.ncbi.nlm.nih.gov/books/NBK321151/ PMID 26447268
- [Background] Dunn K, Bayer LL, Mody SK. Postpartum contraception: An exploratory study of lactation consultants' knowledge and practices. Contraception. 2016 Jul;94(1):87-92. doi: 10.1016/j.contraception.2016.03.007. Epub 2016 Mar 17. PMID 26996737
- [Background] Duvan CI, Gozdemir E, Kaygusuz I, Kamalak Z, Turhan NO. Etonogestrel contraceptive implant (Implanon): analysis of patient compliance and adverse effects in the breastfeeding period. J Turk Ger Gynecol Assoc. 2010 Sep 1;11(3):141-4. doi: 10.5152/jtgga.2010.21. eCollection 2010. PMID 24591920
- [Background] Gurtcheff SE, Turok DK, Stoddard G, Murphy PA, Gibson M, Jones KP. Lactogenesis after early postpartum use of the contraceptive implant: a randomized controlled trial. Obstet Gynecol. 2011 May;117(5):1114-1121. doi: 10.1097/AOG.0b013e3182165ee8. PMID 21508750
- [Background] Taneepanichskul S, Reinprayoon D, Thaithumyanon P, Praisuwanna P, Tosukhowong P, Dieben T. Effects of the etonogestrel-releasing implant Implanon and a nonmedicated intrauterine device on the growth of breast-fed infants. Contraception. 2006 Apr;73(4):368-71. doi: 10.1016/j.contraception.2005.10.010. Epub 2005 Dec 27. PMID 16531169
- [Background] Brito MB, Ferriani RA, Quintana SM, Yazlle ME, Silva de Sa MF, Vieira CS. Safety of the etonogestrel-releasing implant during the immediate postpartum period: a pilot study. Contraception. 2009 Dec;80(6):519-26. doi: 10.1016/j.contraception.2009.05.124. Epub 2009 Jul 10. PMID 19913145
- [Background] Braga GC, Ferriolli E, Quintana SM, Ferriani RA, Pfrimer K, Vieira CS. Immediate postpartum initiation of etonogestrel-releasing implant: A randomized controlled trial on breastfeeding impact. Contraception. 2015 Dec;92(6):536-42. doi: 10.1016/j.contraception.2015.07.009. Epub 2015 Jul 23. PMID 26209863
- [Background] Chapman DJ, Perez-Escamilla R. Maternal perception of the onset of lactation is a valid, public health indicator of lactogenesis stage II. J Nutr. 2000 Dec;130(12):2972-80. doi: 10.1093/jn/130.12.2972. PMID 11110856
- [Background] Sievers E, Haase S, Oldigs HD, Schaub J. The impact of peripartum factors on the onset and duration of lactation. Biol Neonate. 2003;83(4):246-52. doi: 10.1159/000069485. PMID 12743453
- [Background] Dewey KG. Maternal and fetal stress are associated with impaired lactogenesis in humans. J Nutr. 2001 Nov;131(11):3012S-5S. doi: 10.1093/jn/131.11.3012S. PMID 11694638

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Delivery Room Insertion | Postpartum Insertion
Started | 48 | 47
Intent-to-Treat (ITT) Population (ITT population includes participants who were randomized and received the Nexplanon implant) | 38 | 39
Per Protocol Population (Received implant at protocol-specified time point) | 35 | 35
Completed | 35 | 35
Not Completed | 13 | 12

BASELINE CHARACTERISTICS:
Population: Per Protocol Population (received implant at protocol-specified time point)
Groups:
- Total: Total of all reporting groups
Arm/Group | Delivery Room Insertion | Postpartum Insertion | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.7 (5.3) | 26.8 (5.3) | 25.6 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 35 | 70
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 29 | 27 | 56
  Race: Black or African America | 2 | 2 | 4
  Race: Asia | 0 | 2 | 2
  Race: Native American, Hawaiian or Alaskan | 1 | 2 | 3
  Race: Declined to state | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 35 | 35 | 70
Gestational age at delivery (weeks), median (range) [Median (Full Range); unit: weeks] | 39.4 [37 to 41] | 39.1 [33 to 41] | 39.3 [35 to 41]

OUTCOME MEASURES:

1. Primary Outcome: Time to Lactogenesis Stage II [Questionnaire]
Description: Lactogenesis Stage II: The initiation of copious milk secretion as documented by maternal perception.
  To obtain measurement of time to lactogenesis, we will document time at which participants perceive initiation of copious milk secretion using a set of specific validated questions and subtract this by the documented time of delivery.
Time Frame: Participants will be monitored daily by the research staff, in the first seven days postpartum, or until lactogenesis reported, beginning at 24-hours following delivery, to determine time to lactogenesis stage II.
Population: Per Protocol Population (received implant at protocol-specified time point)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Delivery Room Insertion | Postpartum Insertion
Number analyzed (Participants) | 35 | 35
hours | 65 (25.1) | 67.5 (35.8)

2. Secondary Outcome: Number of of Participants Actively Breastfeeding
Description: Exclusive breastfeeding means feedling with breast milk only. Any breast feeding means feeding with breast milk, with water and/or formula.
Time Frame: 2 weeks, 4 weeks, 3 months, 6 months, and 12 months after delivery
Population: Participants with available data for the respective time points are included in the analysis
Measure: Count of Participants; unit: Participants
Groups:
- Delivery Room Insertion: Participants who randomize to this arm will receive the contraceptive Etonogestrel-Immediate implant in the Labor and Delivery room (0-2 hours following delivery).
- Postpartum Insertion: Participants who randomize to this arm will receive the Etonogestrel-Delayed contraceptive implant in the postpartum ward room before discharge (24-48 hours following delivery).
Arm/Group | Delivery Room Insertion | Postpartum Insertion
Number analyzed (Participants) | 26 | 28
Participants
  Exclusive - week 2 | 13 | 16
  Exclusive - week 4: number analyzed (Participants) | 20 | 24
  Exclusive - week 4 | 10 | 8
  Exclusive - month 3: number analyzed (Participants) | 22 | 23
  Exclusive - month 3 | 9 | 6
  Exclusive - month 6: number analyzed (Participants) | 19 | 19
  Exclusive - month 6 | 7 | 3
  Any - week 2 | 25 | 27
  Any - week 4: number analyzed (Participants) | 20 | 24
  Any - week 4 | 17 | 22
  Any - month 3: number analyzed (Participants) | 22 | 23
  Any - month 3 | 18 | 20
  Any - month 6: number analyzed (Participants) | 19 | 19
  Any - month 6 | 13 | 13
  Any - month 12: number analyzed (Participants) | 10 | 13
  Any - month 12 | 5 | 7

3. Secondary Outcome: Number of Participants Still With the Contraceptive Implant at Month 12.
Time Frame: month 12
Population: Participants with available data are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Delivery Room Insertion | Postpartum Insertion
Number analyzed (Participants) | 15 | 14
Participants | 14 | 12

4. Secondary Outcome: Number of Participants Satisfied or Very Satisfied With Implant Contraceptive
Description: Participant-rated as very satisfied, satisfied, neither satisfied or dissatisfied, dissatisfied, or very dissatisfied.
Time Frame: month 12
Population: Participants with available data are included in the analyses
Measure: Count of Participants; unit: Participants
Arm/Group | Delivery Room Insertion | Postpartum Insertion
Number analyzed (Participants) | 18 | 16
Participants | 16 | 10

5. Secondary Outcome: Number of Participants Reporting a Pregnancy Within 12 Months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Delivery Room Insertion | Postpartum Insertion
Number analyzed (Participants) | 35 | 35
Participants | 1 | 1

6. Secondary Outcome: Number of Participants Attending a Postpartum Care Visit by Month 3
Time Frame: month 3
Population: Participants with available data are included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Delivery Room Insertion | Postpartum Insertion
Number analyzed (Participants) | 31 | 29
Participants | 17 | 24

ADVERSE EVENTS:
Time Frame: Time of enrollment through the discharge from the hospital (up to 10 days post-delivery).
Arm/Group | Delivery Room Insertion | Postpartum Insertion
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/47
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/47
Other Adverse Events (participants affected / at risk) | 0/48 | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT02866643/Prot_SAP_000.pdf